CLINICAL TRIAL: NCT04331808
Title: Cohort Multiple Randomized Controlled Trials Open-label of Immune Modulatory Drugs and Other Treatments in COVID-19 Patients - Tocilizumab Trial - CORIMUNO-19 - TOCI (CORIMUNO-TOCI)
Brief Title: CORIMUNO-19 - Tocilizumab Trial - TOCI (CORIMUNO-TOCI)
Acronym: CORIMUNO-TOC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200375-1
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2020-03

CONDITIONS: Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TOCILIZUMAB -- Severe COVID Population (WHO Clinical Progression Scale =5 at baseline) (Experimental): Tocilizumab 8mg/kg on day 1 and if no response (no decrease of oxygen requirement) a second injection at day 3 (fixed dose of 400 mg) CPS: Clinical Progression Scale
  Interventions: Drug: Tocilizumab
- Standard of care -- Severe COVID Population (WHO Clinical Progression Scale =5 at baseline) (No Intervention): Usual care was provided at the discretion of the clinicians
- TOCILIZUMAB -- Critical COVID Population (WHO Clinical Progression Scale >5 at baseline) (Experimental): Tocilizumab 8mg/kg on day 1 and if no response (no decrease of oxygen requirement) a second injection at day 3 (fixed dose of 400 mg) CPS: Clinical Progression Scale
  Interventions: Drug: Tocilizumab
- Standard of care -- Critical COVID Population (WHO Clinical Progression Scale >5 at baseline) (No Intervention): Usual care was provided at the discretion of the clinicians

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab 8mg/kg on day 1 and if no response (no decrease of oxygen requirement) a second injection at day 3 (fixed dose of 400 mg)
  Arms: TOCILIZUMAB -- Critical COVID Population (WHO Clinical Progression Scale >5 at baseline); TOCILIZUMAB -- Severe COVID Population (WHO Clinical Progression Scale =5 at baseline)

SUMMARY:
The overall objective of the study is to determine the therapeutic effect and tolerance of Tocilizumab in patients with moderate, severe pneumonia or critical pneumonia associated with Coronavirus disease 2019 (COVID-19). Tocilizumab (TCZ) is an anti-human IL-6 receptor monoclonal antibody that inhibits signal transduction by binding sIL-6R and mIL-6R. The study has a cohort multiple Randomized Controlled Trials (cmRCT) design. Randomization will occur prior to offering Tocilizumab administration to patients enrolled in the CORIMUNO-19 cohort. Tocilizumab will be administered to consenting adult patients hospitalized with CORVID-19 either diagnosed with moderate or severe pneumonia requiring no mechanical ventilation or critical pneumonia requiring mechanical ventilation. Patients who will chose not to receive Tocilizumab will receive standard of cares. Outcomes of Tocilizumab-treated patients will be compared with outcomes of standard of care treated patients as well as outcomes of patients treated with other immune modulators.

ELIGIBILITY:
Inclusion Criteria:

1. Patients included in the CORIMUNO-19 cohort
2. Patients belonging to one of the 2 following groups:

   * Group 1: Cases meeting all of the following criteria

     * Requiring more than 3L/min of oxygen
     * OMS/WHO progression scale = 5
     * No Non Invasive Ventilation or High flow
   * Group 2: Cases meeting all of the following criteria

     * Respiratory failure AND (requiring mechanical ventilation OR Non Invasive Ventilation OR High flow)
     * WHO progression scale >=6
     * No do-not-resuscitate order (DNR order)

Exclusion Criteria:

* Patients with exclusion criteria to the CORIMUNO-19 cohort.
* Known hypersensitivity to Tocilizumab or to any of their excipients.
* Pregnancy
* Current documented bacterial infection
* Patient with any of following laboratory results out of the ranges detailed below at screening should be discussed depending of the medication:
* Absolute neutrophil count (ANC) ≤ 1.0 x 109/L
* Haemoglobin level: no limitation
* Platelets (PLT) < 50 G /L
* SGOT or SGPT > 5N

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier MARIETTE, MD PhD, Principal Investigator — Hôpital Bicêtre, Assistance Publique-Hôpitaux de Paris
Locations (8):
- France (8):
  - APHP- Hopital Tenon, Paris
  - APHP - Beaujon, Paris
  - APHP - Bichat, Paris
  - APHP - Hopital Necker, Paris
  - APHP - Pitié Salpêtrière, Paris
  - APHP - Saint Louis, Paris
  - CHU Strasbourg, Strasbourg
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Hermine O, Mariette X, Tharaux PL, Resche-Rigon M, Porcher R, Ravaud P; CORIMUNO-19 Collaborative Group. Effect of Tocilizumab vs Usual Care in Adults Hospitalized With COVID-19 and Moderate or Severe Pneumonia: A Randomized Clinical Trial. JAMA Intern Med. 2021 Jan 1;181(1):32-40. doi: 10.1001/jamainternmed.2020.6820. PMID 33080017
- [Result] Mariette X, Hermine O, Tharaux PL, Resche-Rigon M, Steg PG, Porcher R, Ravaud P. Effectiveness of Tocilizumab in Patients Hospitalized With COVID-19: A Follow-up of the CORIMUNO-TOCI-1 Randomized Clinical Trial. JAMA Intern Med. 2021 Sep 1;181(9):1241-1243. doi: 10.1001/jamainternmed.2021.2209. PMID 34028504
- [Result] Hermine O, Mariette X, Porcher R, Resche-Rigon M, Tharaux PL, Ravaud P; CORIMUNO-19 Collaborative Group. Effect of interleukin-6 receptor antagonists in critically ill adult patients with COVID-19 pneumonia: two randomised controlled trials of the CORIMUNO-19 Collaborative Group. Eur Respir J. 2022 Aug 10;60(2):2102523. doi: 10.1183/13993003.02523-2021. Print 2022 Aug. PMID 35115337
- [Derived] Lenoir O, Morin F, Walter-Petrich A, Resmini L, Zaidan M, Mahtal N, Ferlicot S, Puelles VG, Wanner N, Dang J, d'Izarny-Gargas T, Biermann J, Izar B, Baron S, Terrier B, Massy ZA, Essig M, Couturier A, May O, Belenfant X, Buob D, Brocheriou I, Izzedine H, Lombardi Y, Francois H, Moktefi A, Audard V, Sannier A, Daugas E, Jamme M, Henry G, Le Monnier de Gouville I, Marie C, Homyrda L, Verstuyft C, Tubiana S, Kafif O, Piquard V, Dougados M, Huber TB, Livrozet M, Hulot JS, Laouenan C, Ghosn J, Mentre F, Karras A, Yazdanpanah Y, Porcher R, Ravaud P, Caillat-Zucman S, Mariette X, Hermine O, Resche-Rigon M, Tharaux PL; CORIMUNO-19 collaborative group. Levels of circulating kidney injury markers and IL-10 identify non-critically ill patients with COVID-19 at risk of death. JCI Insight. 2026 Jan 23;11(2):e198244. doi: 10.1172/jci.insight.198244. eCollection 2026 Jan 23. PMID 41574613
- [Derived] Joly C, Desjardins D, Porcher R, Pere H, Bruneau T, Zhang Q, Bastard P, Cobat A, Resmini L, Lenoir O, Savale L, Lecuroux C, Verstuyft C, Roque-Afonso AM, Veyer D, Baron G, Resche-Rigon M, Ravaud P, Casanova JL, Le Grand R, Hermine O, Tharaux PL, Mariette X. More rapid blood interferon alpha2 decline in fatal versus surviving COVID-19 patients. Front Immunol. 2023 Nov 21;14:1250214. doi: 10.3389/fimmu.2023.1250214. eCollection 2023. PMID 38077399
- [Derived] Tleyjeh IM. The Misleading "Pooled Effect Estimate" of Crude Data from Observational Studies at Critical Risk of Bias: The Case of Tocilizumab in Coronavirus Disease 2019 (COVID-19). Clin Infect Dis. 2021 Jun 15;72(12):e1154-e1155. doi: 10.1093/cid/ciaa1735. No abstract available. PMID 33201228

RESULTS

PARTICIPANT FLOW:
Groups:
- TOCILIZUMAB -- Severe COVID Population (WHO-CPS =5); TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5): Tocilizumab 8mg/kg on day 1 and if no response (no decrease of oxygen requirement) a second injection at day 3 (fixed dose of 400 mg)
- Standard of Care -- Severe COVID Population (WHO-CPS =5); Standard of Care -- Critical COVID Population (WHO-CPS >5): Usual care was provided at the discretion of the clinicians
Period: Overall Study
Arm/Group | TOCILIZUMAB -- Severe COVID Population (WHO-CPS =5) | Standard of Care -- Severe COVID Population (WHO-CPS =5) | TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5)
Started | 64 | 67 | 51 | 46
Completed | 63 | 67 | 49 | 43
Not Completed | 1 | 0 | 2 | 3
Not completed — Withdrew consent | 1 | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TOCILIZUMAB -- Severe COVID Population (WHO-CPS =5) | Standard of Care -- Severe COVID Population (WHO-CPS =5) | TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5) | Total
Number analyzed (Participants) | 63 | 67 | 49 | 43 | 222
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [57.1 to 74.3] | 63.3 [57.1 to 72.3] | 63.2 [59.4 to 70.9] | 65.4 [57.6 to 70.5] | 64 [57.3 to 71.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 23 | 16 | 10 | 68
  Male | 44 | 44 | 33 | 33 | 154
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m²] — kg/m² Population: Missing data are possible
  kg/m²
    number analyzed (Participants) | 46 | 46 | 47 | 37 | 176
    (all) | 27.9 [23.3 to 30.8] | 27.4 [24.5 to 31.3] | 27.8 [24.8 to 31.4] | 28.7 [25.4 to 31.6] | 27.8 [24.6 to 31.3]
Weight [Median (Inter-Quartile Range); unit: kg] — Population: Missing data are possible
  kg
    number analyzed (Participants) | 63 | 55 | 49 | 40 | 207
    (all) | 80 [70 to 90] | 78 [70 to 90] | 80 [70 to 95] | 81 [75 to 90.5] | 80 [70 to 92]
SPO2 [Median (Inter-Quartile Range); unit: %] — Population: Missing data are possible
  %
    number analyzed (Participants) | 63 | 67 | 48 | 43 | 221
    (all) | 95 [93 to 96] | 95 [93 to 97] | 94 [92 to 96] | 91 [91 to 98] | 95 [93 to 97]
Temperature [Median (Inter-Quartile Range); unit: °c] | 37.3 [36.8 to 38.2] | 37.9 [37 to 38.6] | 37.7 [37 to 38.6] | 38 [37 to 38.7] | 37.7 [37 to 38.5]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With WHO Clinical Progression Scale > 5 at Day 4 -- Severe COVID Population (WHO Clinical Progression Scale =5 at Baseline)
Description: Percentage of participants who has died or needed non-invasive or mechanical ventilation by day 4 (WHO clinical progression scale > 5). A patient with new do-not-resuscitate order at day 4 will be considered as with a score > 5.
  WHO progression scale:
  Uninfected; non viral RNA detected: 0 Asymptomatic; viral RNA detected: 1 Symptomatic; Independent: 2 Symptomatic; Assistance needed: 3 Hospitalized; No oxygen therapy: 4 Hospitalized; oxygen by mask or nasal prongs: 5 Hospitalized; oxygen by NIV or High flow: 6 Intubation and Mechanical ventilation, pO2/FIO2>=150 OR SpO2/FIO2>=200: 7 Mechanical ventilation, (pO2/FIO2<150 OR SpO2/FIO2<200) OR vasopressors (norepinephrine >0.3 microg/kg/min): 8 Mechanical ventilation, pO2/FIO2<150 AND vasopressors (norepinephrine >0.3 microg/kg/min), OR Dialysis OR ECMO: 9 Dead: 10
Time Frame: 4 days
Population: Severe COVID Population (WHO clinical progression scale =5 at baseline)
Measure: Number; unit: percentage of participants
Arm/Group | TOCILIZUMAB -- Severe COVID Population (WHO-CPS =5) | Standard of Care -- Severe COVID Population (WHO-CPS =5)
Number analyzed (Participants) | 64 | 67
percentage of participants | 19 | 28
Statistical Analysis 1: Comparison: TOCILIZUMAB -- Severe COVID Population (WHO-CPS =5) vs Standard of Care -- Severe COVID Population (WHO-CPS =5); Test type: Superiority; Bayesian analysis — Posterior probability; Adjusted for age and centre; Median posterior absolute risk differenc = -9, 90% CI 2-sided [-21.0 to 3.1] — % Confidence Interval is % Credibility interval here

2. Primary Outcome: Percentage of Participants With Non-invasive Ventilation, Mechanical Ventilation or Death at Day 14 (WHO Clinical Progression Scale =5 at Baseline)
Description: Survival without needs of ventilator utilization (including non invasive ventilation and high flow) at day 14. Percentage of non-invasive ventilation, mechanical ventilation or death. Thus, events considered are needing ventilator utilization (mechanical or non-invasive ventilation including high flow oxygen), or death. New do-not-resuscitate (DNR) order (if given after the inclusion of the patient) will be considered as an event at the date of the DNR.
Time Frame: Day 1 to Day 14
Population: Severe COVID Population (WHO clinical progression scale =5 at baseline)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TOCILIZUMAB -- Severe COVID Population (WHO-CPS =5) | Standard of Care -- Severe COVID Population (WHO-CPS =5)
Number analyzed (Participants) | 49 | 43
percentage of participants | 24 [13 to 34] | 36 [23 to 46]
Statistical Analysis 1: Comparison: TOCILIZUMAB -- Severe COVID Population (WHO-CPS =5) vs Standard of Care -- Severe COVID Population (WHO-CPS =5); Test type: Superiority; Bayesian analysis — Posterior probability; HR adjusted for age and centre; Median posterior Hazard Ratio = 0.58, 90% CI 2-sided [0.33 to 1.00] — % Confidence interval is % Credible Interval here

3. Primary Outcome: Percentage of Participants With no Improvement in WHO Clinical Progression Scale at Day 4 -- Critical COVID Population ( WHO Clinical Progression Scale >5 at Baseline)
Description: Results are presented as the percentage not improved, so that an effective treatment would be associated with a decrease in percentage
  WHO progression scale:
  Uninfected; non viral RNA detected: 0 Asymptomatic; viral RNA detected: 1 Symptomatic; Independent: 2 Symptomatic; Assistance needed: 3 Hospitalized; No oxygen therapy: 4 Hospitalized; oxygen by mask or nasal prongs: 5 Hospitalized; oxygen by NIV or High flow: 6 Intubation and Mechanical ventilation, pO2/FIO2>=150 OR SpO2/FIO2>=200: 7 Mechanical ventilation, (pO2/FIO2<150 OR SpO2/FIO2<200) OR vasopressors (norepinephrine >0.3 microg/kg/min): 8 Mechanical ventilation, pO2/FIO2<150 AND vasopressors (norepinephrine >0.3 microg/kg/min), OR Dialysis OR ECMO: 9 Dead: 10
Time Frame: 4 days
Population: Critical COVID population ( WHO Clinical Progression Scale >5 at baseline)
Measure: Number; unit: percentage of participants
Arm/Group | TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5)
Number analyzed (Participants) | 49 | 43
percentage of participants | 71 | 70
Statistical Analysis 1: Comparison: TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Test type: Superiority; Bayesian analysis — Posterior probability; Adjusted for age and centre; Median posterior absolute risk differenc = 1.7, 90% CI 2-sided [-13.6 to 17.1] — % Confidence Interval is % Credible Interval here Results are presented as the proportion not improved, so that an effective treatment would be associated with a decrease in proportion

4. Primary Outcome: Cumulative Incidence (Percentage of Participants) With Successful Tracheal Extubation at Day 14 -- Critical COVID Population (WHO Clinical Progression Scale >5 at Baseline)
Description: Cumulative incidence of successful tracheal extubation (defined as duration extubation > 48h) at day 14 if patients have been intubated before day 14 ; or removal of Non Invasive Ventilation or high flow (for > 48h) if they were included under oxygen by Non Invasive Ventilation or High flow (score 6) and remained without intubation. Death or new do-not-resuscitate order (if given after the inclusion of the patient) will be considered as a competing event.
Time Frame: Day 1 to Day 14
Population: Critical COVID Population (WHO clinical progression scale >5 at baseline)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5)
Number analyzed (Participants) | 49 | 43
percentage of participants | 47 [32 to 60] | 42 [27 to 56]
Statistical Analysis 1: Comparison: TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Test type: Superiority; Bayesian analysis — Posterior probability; HR adjusted for age and centre; Median posterior Hazard Ratio = 1.19, 90% CI 2-sided [0.71 to 2.04] — % Confidence interval is % Credible Interval here

5. Secondary Outcome: Percentage of Participants Surviving (Overall Survival)
Description: Percentage of participants surviving at 14, 28 and 90 days
Time Frame: 14, 28 and 90 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TOCILIZUMAB -- Severe COVID Population (WHO-CPS =5) | Standard of Care -- Severe COVID Population (WHO-CPS =5) | TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5)
Number analyzed (Participants) | 63 | 67 | 49 | 43
percentage of participants
  Day 14 | 89 [81 to 97] | 91 [84 to 98] | 90 [82 to 99] | 79 [68 to 92]
  Day 28 | 89 [81 to 97] | 88 [80 to 96] | 84 [74 to 95] | 77 [65 to 90]
  Day 90 | 89 [81 to 97] | 84 [75 to 93] | 76 [64 to 89] | 70 [57 to 85]
Statistical Analysis 1: Comparison: TOCILIZUMAB -- Severe COVID Population (WHO-CPS =5) vs Standard of Care -- Severe COVID Population (WHO-CPS =5); Day 14; Test type: Superiority; Regression, Cox; adjusted for age and sex; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.40 to 3.55]
Statistical Analysis 2: Comparison: TOCILIZUMAB -- Severe COVID Population (WHO-CPS =5) vs Standard of Care -- Severe COVID Population (WHO-CPS =5); Day 28; Test type: Superiority; Regression, Cox; adjusted for age and centre; Cox Proportional Hazard = 0.92, 95% CI 2-sided [0.33 to 2.53]
Statistical Analysis 3: Comparison: TOCILIZUMAB -- Severe COVID Population (WHO-CPS =5) vs Standard of Care -- Severe COVID Population (WHO-CPS =5); Day 90; Test type: Superiority; Regression, Cox; adjusted for age and centre; Cox Proportional Hazard = 0.64, 95% CI 2-sided [0.25 to 1.65]
Statistical Analysis 4: Comparison: TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Day 14; Test type: Superiority; Regression, Cox; adjusted for age and centre; Hazard Ratio (HR) = 0.37, 95% CI 2-sided [0.12 to 1.15]
Statistical Analysis 5: Comparison: TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Day 28; Test type: Superiority; Regression, Cox; adjusted for age and centre; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.32 to 1.47]
Statistical Analysis 6: Comparison: TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Day 90; Test type: Superiority; Regression, Cox; adjusted for age and centre; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.30 to 1.49]

6. Secondary Outcome: WHO Progression Scale
Description: WHO progression scale:
  Uninfected; non viral RNA detected: 0 Asymptomatic; viral RNA detected: 1 Symptomatic; Independent: 2 Symptomatic; Assistance needed: 3 Hospitalized; No oxygen therapy: 4 Hospitalized; oxygen by mask or nasal prongs: 5 Hospitalized; oxygen by NIV or High flow: 6 Intubation and Mechanical ventilation, pO2/FIO2>=150 OR SpO2/FIO2>=200: 7 Mechanical ventilation, (pO2/FIO2<150 OR SpO2/FIO2<200) OR vasopressors (norepinephrine >0.3 microg/kg/min): 8 Mechanical ventilation, pO2/FIO2<150 AND vasopressors (norepinephrine >0.3 microg/kg/min), OR Dialysis OR ECMO: 9 Dead: 10
Time Frame: 4, 7 and 14 days
Population: Missing data are possible
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | TOCILIZUMAB -- Severe COVID Population (WHO-CPS =5) | Standard of Care -- Severe COVID Population (WHO-CPS =5) | TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5)
Number analyzed (Participants) | 63 | 67 | 49 | 43
units on a scale
  Day 4 | 5 [5 to 5] | 5 [5 to 6] | 7 [7 to 8] | 8 [7 to 8]
  Day 7: number analyzed (Participants) | 55 | 64 | 48 | 43
  Day 7 | 5 [5 to 5] | 5 [5 to 6] | 7 [5 to 8] | 8 [7 to 8]
  Day 14: number analyzed (Participants) | 59 | 65 | 48 | 43
  Day 14 | 2 [2 to 5] | 4 [2 to 7] | 7 [5 to 8] | 7 [5 to 9]
Statistical Analysis 1: Comparison: TOCILIZUMAB -- Severe COVID Population (WHO-CPS =5) vs Standard of Care -- Severe COVID Population (WHO-CPS =5); Day 4; Test type: Superiority; Proportionnal odds model; Bayesian analysis. Adjusted for age and centre; Median posterior OR = 0.60, 95% CI 2-sided [0.27 to 1.28] — % Confidence Interval is % Credible Interval here
Statistical Analysis 2: Comparison: TOCILIZUMAB -- Severe COVID Population (WHO-CPS =5) vs Standard of Care -- Severe COVID Population (WHO-CPS =5); Day 7; Test type: Superiority; Proportionnal odds model; Bayesian analysis. Adjusted for age and centre; Median posterior OR = 0.86, 95% CI 2-sided [0.43 to 1.71]; % Confidence Interval is % Credible Interval here
Statistical Analysis 3: Comparison: TOCILIZUMAB -- Severe COVID Population (WHO-CPS =5) vs Standard of Care -- Severe COVID Population (WHO-CPS =5); Day 14; Test type: Superiority; Proportionnal odds model; Bayesian analysis. Adjusted for age and sex; Median posterior OR = 0.76, 95% CI 2-sided [0.40 to 1.42] — % Confidence Interval is % Credible Interval here
Statistical Analysis 4: Comparison: TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Day 4; Test type: Superiority; Proportionnal odds model; Bayesian analysis. Adjusted for age and centre; Median posterior OR = 0.85, 95% CI 2-sided [0.39 to 1.82]; % Confidence Interval is % Credible Interval here
Statistical Analysis 5: Comparison: TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Day 7; Test type: Superiority; Proportionnal odds model; Bayesian analysis. Adjusted for age and centre; Median posterior OR = 0.69, 95% CI 2-sided [0.32 to 1.47] — % Confidence Interval is % Credible Interval here
Statistical Analysis 6: Comparison: TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Day 14; Test type: Superiority; Proportionnal odds model; Bayesian analysis. Adjusted for age and centre; Median posterior OR = 0.68, 95% CI 2-sided [0.32 to 1.43] — % Confidence Interval is % Credible Interval here

7. Secondary Outcome: Mean of Ventilator Free-days at Day 28 -- Critical COVID Population (WHO-clinical Progression Scale >5 at Baseline)
Description: 28-day ventilator free-days
Time Frame: 28 days
Population: Critical COVID Population (WHO clinical progression scale >5 at baseline)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5)
Number analyzed (Participants) | 49 | 43
days | 12.8 (10.7) | 10.3 (11.1)
Statistical Analysis 1: Comparison: TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Test type: Superiority; adjusted on age and centre; Mean Difference (Net) = -2.5, 95% CI 2-sided [-6.9 to 1.7]

8. Secondary Outcome: Cumulative Incidence (Percentage of Participants) of Oxygen Supply Independency
Description: Time to oxygen supply independency
Time Frame: Day 28, 90
Population: No assessment in Severe COVID Population (WHO Clinical Progression Scale =5 at baseline) at Day 90
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TOCILIZUMAB -- Severe COVID Population (WHO-CPS =5) | Standard of Care -- Severe COVID Population (WHO-CPS =5) | TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5)
Number analyzed (Participants) | 63 | 67 | 49 | 43
percentage of participants
  Day 28 | 89 [78 to 95] | 75 [62 to 83] | 59 [44 to 72] | 49 [33 to 63]
  Day 90: number analyzed (Participants) | 0 | 0 | 49 | 43
  Day 90 |  |  | 69 [53 to 80] | 64 [47 to 77]
Statistical Analysis 1: Comparison: TOCILIZUMAB -- Severe COVID Population (WHO-CPS =5) vs Standard of Care -- Severe COVID Population (WHO-CPS =5); Day 28; Test type: Superiority; Fine-Gray model; adjusted for age and centre; Hazard Ratio (HR) = 1.41, 95% CI 2-sided [0.98 to 2.01]
Statistical Analysis 2: Comparison: TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Day 28; Test type: Superiority; Fine-Gray model; Hazard Ratio (HR) = 1.44, 95% CI 2-sided [0.82 to 2.52]
Statistical Analysis 3: Comparison: TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Day 90; Test type: Superiority; Fine-Gray model; adjusted on age and centre; Hazard Ratio (HR) = 1.28, 95% CI 2-sided [0.80 to 2.03]

9. Secondary Outcome: Cumulative Incidence (Percentage of Participants) of Discharge From Hospital
Description: Time to discharge from hospital
Time Frame: 28, 90 days
Population: No assessment in Severe COVID Population (WHO Clinical Progression Scale =5 at baseline) at Day 90
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TOCILIZUMAB -- Severe COVID Population (WHO-CPS =5) | Standard of Care -- Severe COVID Population (WHO-CPS =5) | TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5)
Number analyzed (Participants) | 63 | 67 | 49 | 43
percentage of participants
  Day 28 | 83 [70 to 90] | 73 [61 to 82] | 55 [40 to 68] | 42 [27 to 56]
  Day 90: number analyzed (Participants) | 0 | 0 | 49 | 43
  Day 90 |  |  | 70 [54 to 82] | 60 [44 to 74]
Statistical Analysis 1: Comparison: TOCILIZUMAB -- Severe COVID Population (WHO-CPS =5) vs Standard of Care -- Severe COVID Population (WHO-CPS =5); Day 28; Test type: Superiority; Fine-Gray model; adjusted on age and centre; Hazard Ratio (HR) = 1.52, 95% CI 2-sided [1.02 to 2.27]
Statistical Analysis 2: Comparison: TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Day 28; Test type: Superiority; Fine-Gray model; adjusted for age and centre; Hazard Ratio (HR) = 1.45, 95% CI 2-sided [0.80 to 2.63]
Statistical Analysis 3: Comparison: TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Day 90; Test type: Superiority; Fine-Gray model; adjusted for age and centre; Hazard Ratio (HR) = 1.35, 95% CI 2-sided [0.84 to 2.17]

10. Secondary Outcome: Cumulative Incidence (Percentage of Participants) of Intensive Care Unit Discharge -- Critical COVID Population (WHO Clinical Progression Scale >5 at Baseline)
Description: Time to discharge from Intensive Care Unit
Time Frame: 28, 90 days
Population: Critical COVID Population (WHO clinical progression scale >5 at baseline) Patients in intensive care unit at inclusion
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5)
Number analyzed (Participants) | 40 | 37
percentage of participants
  Day 28 | 72 [55 to 84] | 60 [42 to 74]
  Day 90 | 84 [66 to 93] | 83 [63 to 93]
Statistical Analysis 1: Comparison: TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Day 28; Test type: Superiority; Fine-Gray model; adjusted on age and centre; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.73 to 1.81]
Statistical Analysis 2: Comparison: TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Day 90; Test type: Superiority; Fine-Gray model; adjusted on age and centre; Hazard Ratio (HR) = 1.28, 95% CI 2-sided [0.73 to 2.24]

11. Secondary Outcome: PaO2/FIO2 Ratio -- Critical COVID Population (WHO Clinical Progression Scale >5 at Baseline)
Description: Evolution of PaO2/FiO2 ratio PaO2 is partial pressure of arterial oxygen expressed in mmHg. FiO2 is fraction of inspired oxygen (for instance, 0.33 for 33% oxygen) with no units.
  PaO2/FiO2 ratio is expressed in mmHg.
Time Frame: day 1 to day 14
Population: No statistical comparison was performed due to the limited number of patients with available follow-up data.
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5)
Number analyzed (Participants) | 36 | 30
mmHg
  Day 1: number analyzed (Participants) | 36 | 28
  Day 1 | 155.1 [98.4 to 201.8] | 135.0 [98.8 to 184.7]
  Day 4: number analyzed (Participants) | 33 | 30
  Day 4 | 144.0 [95.7 to 214.0] | 143.8 [96.2 to 175.2]
  Day7: number analyzed (Participants) | 27 | 22
  Day7 | 126.0 [89.7 to 190.0] | 142.8 [105.5 to 199.0]
  Day 14: number analyzed (Participants) | 8 | 6
  Day 14 | 153.7 [141.2 to 189.5] | 94.0 [86.2 to 129.5]

ADVERSE EVENTS:
Time Frame: Adverse events were systematically assessed at Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13 and 14 while participants were inpatient, and at Days 28 and 60 and 90.
Description: Only deaths and serious adverse events were reported. "0" total Number of Participants at Risk means " Other (Not Including Serious) Adverse Events were not monitored/analyzed ".
Arm/Group | TOCILIZUMAB -- Severe COVID Population (WHO-CPS =5) | Standard of Care -- Severe COVID Population (WHO-CPS =5) | TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5)
All-Cause Mortality (participants affected / at risk) | 7/63 | 11/67 | 12/49 | 13/43
Serious Adverse Events (participants affected / at risk) | 20/63 | 29/67 | 31/49 | 27/43
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TOCILIZUMAB -- Severe COVID Population (WHO-CPS =5) (N=63) | Standard of Care -- Severe COVID Population (WHO-CPS =5) (N=67) | TOCILIZUMAB -- Critical COVID Population (WHO-CPS >5) (N=49) | Standard of Care -- Critical COVID Population (WHO-CPS >5) (N=43)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anemia (General disorders) | 1 (1) | 4 (4) | 6 (7) | 7 (7)
Hyperlipasemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Hepatic cytolysis (Hepatobiliary disorders) | 4 (4) | 3 (4) | 8 (9) | 3 (3)
Multiple organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Vascular disorders) | 0 (0) | 3 (3) | 4 (4) | 1 (1)
Fever (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperkaliemia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 2 (2) | 4 (4) | 3 (4)
Arterial ischemia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 16 (19) | 10 (13) | 13 (15)
Bacterial sepsis (Infections and infestations) | 1 (2) | 8 (11) | 10 (25) | 7 (12)
Fungal sepsis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Viral sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tetraparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Ischemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypovolemic shock (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Severe acute pancreatis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperleukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arterial hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Guillain Barré syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bleeding (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb ischemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tracheotomy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Psoas hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT04331808/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-13): https://cdn.clinicaltrials.gov/large-docs/08/NCT04331808/SAP_001.pdf